CLINICAL TRIAL: NCT06583356
Title: The Adaptation and Effectiveness of Motivational Interviewing Intervention For Risky Drinking Treatment Among Indigenous Population: Protocol For A Single-arm Trial
Brief Title: Motivational Interviewing Intervention For Risky Drinking Treatment Among Indigenous Population
Acronym: MIRDIP
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Department of Public Health Medicine, MARA University of Technology (Other)
Responsible Party: Principal Investigator, Rifhan Rasuli, Doctor of Public Health student, Department of Public Health Medicine, MARA University of Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RSCH ID-24-01486-I7A
Record Dates: First submitted 2024-09-01; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Alcohol Abuse
Keywords: motivational interviewing, risky drinking
MeSH Terms: conditions — Alcoholism | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Motivational interviewing (Experimental): Will receive motivational interviewing intervention previously, delivered face-to-face at participants' home, 1 session, followed by 2 brief follow-up sessions. Each session is expected to last approximately 30 to 45 minutes.
  Interventions: Behavioral: Motivational interviewing

INTERVENTIONS:
Behavioral: Motivational interviewing — Participants will receive motivational interviewing intervention previously, delivered face-to-face at participants' home, 1 session, followed by 2 brief follow-up sessions. Each session is expected to last approximately 30 to 45 minutes.

SUMMARY:
The goal of this single-arm trial is to adapt and evaluate the effectiveness of motivational interviewing intervention for treating risky drinking behaviour among indigenous population in Pahang, Malaysia.

To achieve this, the investigators will:

i) Translate 3 questionnaires regarding alcohol consumption from English into Jakun language (a language of one of Malaysia&#39;s indigenous communities) ii) Adapt a motivational interviewing intervention for treatment of risky drinking for this community iii) Implement the intervention and measure its outcomes using the translated questionnaires

Participants will:

i) Answer translated questionnaires during the validation of questionnaires (phase 1) ii) Receive 3 sessions of motivational interviewing (phase 2)

DETAILED DESCRIPTION:
Alcohol consumption, particularly in the form of harmful alcohol use, has long posed substantial public health challenges. It has been proven to cause multitude health problems, including non-communicable diseases, injuries, and increased risk of communicable diseases (Rehm et al., 2017; Room et al., 2005). Globally, it is estimated there are 2.6 million deaths annually as a result of the harmful alcohol use (WHO, 2024).

Risky drinking is defined as the level of alcohol consumption that is associated with negative consequences, such as health problems, accidents, and social issues (Karlsson et al., 2023). It is defined as Alcohol Use Disorders Identification Test (AUDIT-10) score of more or equal to 8 (Institute for Public Health, 2020; O'Donnell et al., 2018).

Indigenous community in the Peninsular Malaysia is a member of an aboriginal ethnic group who speaks an aboriginal language and habitually follows an aboriginal way of life, customs, and beliefs (Malaysian government, 1954). Among this community, alcohol consumption has long been associated with a tradition during festivals or after a good harvest season (Ali et al., 1991). Nevertheless, studies have found that the prevalence of alcohol consumption among indigenous populations in Malaysia varies from as low as 7.1% to as high as 34.8% (Ahmad et al., 2013; Chua et al., 2017; Ithnin et al., 2020; Yusof et al., 2007), with the most consumed alcohol beverage is beer (Abd Rashid et al., 2010).

Globally, while indigenous populations are more likely to abstain from alcohol, they are more likely to progress to risky drinking, resulting in alcohol-related health consequences (Andersen et al., 2021; Delker et al., 2016; Gray et al., 2018). Possible reasons may include socioeconomic disparities, perceived discrimination and marginalisation (Camacho-Martínez et al., 2023), cultural disconnection (Werito & Belone, 2021), community and social factors (Conigrave et al., 2021), and a lack of access to culturally sensitive health services (Kelaher et al., 2012). Furthermore, a study in Malaysia revealed that alcohol consumption among the indigenous community was primarily driven by stress management strategy and social factors (Ithnina et al., 2020).

There are several approaches in risky drinking intervention, namely pharmacological, psychological, and social support (d&#39;Abbs et al., 2013). Psychological intervention is found to be the most active and studied approach among indigenous populations (d'Abbs et al., 2013; Purcell-Khodr et al., 2020). This includes brief intervention, motivational interviewing, and cognitive behavioural therapy (Andersen et al., 2021; d'Abbs et al., 2013; Purcell-Khodr et al., 2020).

Motivational interviewing is a counselling method to enhance motivation through resolution of ambivalence (Hall et al., 2012). It is a client-oriented counselling style (Miller & Rollnick, 2012), emphasising on a collaborative and non-confrontational approach (Hettema et al., 2005).

Presently, the only available psychological intervention on risky drinking in Malaysia is predominantly based on standard brief intervention designed for the general population, which prioritises imparting information and telling patients what to do. In addition, there is a lack of evaluation on the effectiveness of alcohol psychological intervention among indigenous populations in Malaysia, especially those that are tailored to their cultural and environmental context. Therefore, there is a need to adapt an intervention grounded in motivational interviewing and its effectiveness be tested to address the issue of risky drinking among these populations.

The objective of this study is to adapt and evaluate the effectiveness of MI intervention for treating risky drinking behaviour among indigenous population in the state of Pahang, Malaysia.

This study will be divided into 2 phases:

i) Phase 1, which consists of the translation and validation of questionnaires, and the development of motivational interviewing intervention for risky drinking treatment ii) Phase 2, the single-arm trial

Phase 1 (translation and validation of questionnaires)

Several questionnaires regarding the trial outcomes will need to be translated from English into Jakun, the language of the indigenous tribe where the trial will take place.

Questionnaires to be translated and validated are: i) Readiness to Change Questionnaire (Revised Version) (RCQ); ii) Motivation Thought Frequency Scales for Alcohol (MTF-A); iii) Brief Alcohol Abstinence Self-Efficacy 12-Item (AASE) Scale.

The process of translation and backtranslation are performed by 2 medical experts and 2 language experts. The selection of 2 medical experts is performed using purposive sampling: medical professionals of Jakun origin with experience working in Rompin district, Pahang, Malaysia. The selection of 2 language experts is performed using purposive sampling as well: individuals of Jakun descent in Rompin district who are well-versed in both English and Jakun language, but not knowledgeable about medical terminology.

The harmonised version will undergo face validation among respondents who are selected randomly from RPS Kedaik, the site for the questionnaire validation.

Method to select participants for face validation: From the spot map of the settlement, numbers will be assigned to each house. Simple random sampling will be performed using computer-generated random numbers. A representative from the selected house will be invited to be a respondent.

The resulting finalised version of RCQ-JK, MTF-A-JK, and AASE-JK will undergo a reliability and validation study. From the spot map of the settlement, numbers will be assigned to each house. Simple random sampling will be performed using computer-generated random numbers. A representative from the selected house will be screened i.e. age ≥ 18 years old who is a current drinker. Those who fulfill these criteria will be invited to join the study.

During informed consent process, individual will be briefed using the simple Malay language, with patient information sheet, which is available in Jakun language, as the guide to ensure understanding. Individuals who cannot read can be represented by reliable kin or legally authorised representative.

Phase 1 (adaptation of motivational interviewing intervention for risky drinking treatment)

This process will be guided by ADDIE Model (analysis, design, development, implementation, and evaluation).

In analysis phase, a literature review will be conducted from which evidence are collected to inform the content development process e.g. published articles, manuals, guidelines.

In design phase, findings from the previous literature review will be discussed with a panel of experts using Nominal Group Technique. There will be 4 experts, selected using purposive sampling, which include a public health medicine specialist, a psychologist with certificate in motivational interviewing, a researcher specialised in health promotion, and a medical assistant in the local health clinic who is of Jakun descent. The facilitator (primary investigator) will summarise the scores to ascertain the overall group priorities.

In development phase, the content derived from the previous 2 phases will be developed into a module for motivational interviewing intervention.

At the end of content development, content validity will be assessed by obtaining ratings from each member of the expert panel with regards to its relevance, clarity, simplicity, and ambiguity. Additionally, there would also be content and face validation by another panel of expert.

Implementation and evaluation phases will be conducted during the subsequent single-arm trial.

Phase 2 (single-arm trial)

This trial will be conducted at another indigenous settlement located close to the one in previous phase, called Kampung Jemeri.

Sampling methods: From the spot map of the settlement, numbers will be assigned to each house. Simple random sampling will be performed using computer-generated random numbers. A representative from the selected house will be approached and explained about the study.

During informed consent process, individual will be briefed using simple Malay language, with patient information sheet, which is available in Bahasa Jakun, as the guide to ensure understanding. Individuals who cannot read can be represented by reliable kin or legally authorised representative. If the individual agrees, he/she will be screened using AUDIT-10 questionnaire. Those with AUDIT-10 score between 8 and 19 will subjected to further eligibility criteria (refer inclusion and exclusion criteria for Phase 2). Those who fulfill these criteria will be invited to join the study. Those who do not fulfill these criteria will be thanked and will not be enrolled in the study.

Measurement and data collection Participants' information will be collected at 1st visit, right after 1st intervention, 6 weeks post-intervention, and 3 months post-intervention.

Why measurement is performed at immediately after 1st intervention, 6 weeks and 3 months post-intervention: A systematic review of reviews by Frost et al. (2018) revealed consistent evidence on beneficial effect of motivational interview on alcohol consumption for short term outcomes (less than 4 months), but less consistent evidence on sustained (more than 4 months) outcomes. Furthermore, a systematic review and meta-analysis by Lundahl et al. (2018) measuring the effect size of motivational interviewing indicated that between immediate and 1 month time frame after intervention, MI impact shows odds ratio of 1.38. Between 5 weeks to 6 months, odds ratio increases to 1.72. The odds ratio drops to 1.34 after 7 to 12 months of intervention aspect of the follow-up process.

Strategies to increase participant retention include telephone contact to participants and In-person visits to participants' homes. Given that the follow-up will be conducted face-to-face, reaching the participants at their residences is essentially crucial

Sample size calculation For face validation, the sample size would be 10. Based on Sousa & Rojjanasrirat (2011) who recommended a sample size of 10 to 40 for a pilot testing during the translation, adaptation, and validation of instruments for use in cross-cultural health care research.

For assessment of reliability (internal consistency - Cronbach's alpha) and construct validity (exploratory factor analysis (EFA)), a sample size of 200 will be used.

This recommendation is based on the work of Mokkink et al. (2019), which suggests that for assessing internal consistency, a minimum sample size of 100 is recommended. For factor analysis, the guideline is to have at least 7 times the number of items, with a minimum sample size of 100. Given that each questionnaire has 12 items, the ideal sample size would be 12 items × 7 = 84. However, since 100 is the minimum requirement, the larger sample size of 100 should be used for both internal consistency and factor analysis.

However, to achieve more reliable results, MacCallum et al. (1999) suggested a larger sample between 100 and 200 in case of communalities around 0.5. Hence a sample size of 200 will be used.

For further assessment of construct validity (confirmatory factor analysis (CFA)), a further sample size of 300 will be used. This is based on Mokkink et al. (2019), which proposes 7 times number of items for factor analysis with minimum 100. However, to achieve more reliable results, MacCallum et al. (1999) suggested a larger sample of 300 in case of low communalities.

For the Phase 2 (single-arm trial), the sample size calculation is performed using the equation from paired or matched groups for clinical studies (Machin et al., 2011).

A study by Zatzick et al.(Zatzick et al., 2014) noted reduction of 1.8 (95% CI 1.1, 2.4) in AUDIT-10 score after 6 months following an MI intervention on 409 subjects.

To calculate the standard deviation, CI = 1.96 x Standard error, SE 1.8 - 1.1 = 1.96 x SE SE = 0.357 SE = SD / (√Sample size) 0.357 = SD / (√409) Standard deviation, SD = 0.357 x √409 = 7.22

Width of 95% CI, ω = 2.4 - 1.1 = 1.3 Anticipated standard deviation, σPlan = 7.22 ΛPlan = ω / σPlan = 1.3 / 1.8 = 0.722

Subsequently, the sample size calculation is performed using the above equation, yielding a sample size of 29.48, which is rounded to 30.

This is further confirmed by the table proposed by Machin et al.(Machin et al., 2011). Where ΛPlan between 0.70 and 0.75, which gives m at 95% confidence interval between 55 and 63. When NPairs = m/2, the sample size would be between 27.5 and 31.5.

Accounting for risk for lost to follow-up, additional 20% will be recruited, based on previous studies (Gaume et al., 2022; Jayaraj et al., 2012). Therefore, the minimum sample size would be 36.

Exit strategy:

Any participant who is found to have any of the following condition, will require proper referral to the relevant medical personnel e.g. psychiatrist, hospital: i) Serious mental illness previously undiagnosed; ii) Suspected to have alcohol dependence, as evidence by AUDIT-10 score ≥ 20; iii) Any serious adverse event such as one that is life-threatening or require hospitalisation; iv) Inability to continue participating in the study due to medical reason

Ethical consideration This study requires approval from the Faculty Ethics Review Committee, Faculty of Medicine, MARA University of Technology (UiTM) Malaysia and registration with National Medical Research Register (NMRR), Malaysia. Permission from the Department of Indigenous People Development (JAKOA) is also required. Data collection will only be initiated once the above approvals are obtained.

Informed consent process will be conducted prior to inclusion, using simple Malay language, with patient information sheet, which is available in Bahasa Jakun, as the guide, ensuring that individuals are provided with comprehensive information about the study. Participants will be informed that their involvement is voluntary, and they have the right to withdraw from the study at any time without repercussion.

The counseling session will be conducted one-on-one in a designated area within the participant's home to ensure privacy.

ELIGIBILITY:
Phase 1 (validation of translated questionnaires)

Inclusion Criteria:

* Individuals in the selected settlement age ≥ 18 years old who are current drinkers, irrespective of volume (current drinker is defined as individual who has consumed any alcoholic beverage in the past 12 months)
* Agrees to participate in the study after explanation given

Exclusion Criteria:

* Those with history of serious mental illness or cognitive impairment
* Those who are unable to speak proficient Malay or Jakun language

Phase 2 (single-arm trial):

Inclusion Criteria:

* Individuals in the selected settlement and its surrounding, age ≥ 18 years old who are current drinkers
* Agrees to participate in the study after explanation given

Exclusion Criteria:

* AUDIT-10 score < 8 or > 19
* Those with history of serious mental illness or cognitive impairment
* Those who are currently on other alcohol intervention programmes
* Those who are unable to speak proficient Malay or English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Severity of alcohol consumption | 4 months
  The extent of alcohol-related consequences e.g. social, legal, physical, and psychological problems (Babor et al., 2001). Measured by Alcohol Use Disorders Identification Test (AUDIT-10) score (validated Malay version - already available). Higher AUDIT-10 score indicates more severe alcohol consumption.

SECONDARY OUTCOMES:
Readiness to change | 4 months
  The extent to which an individual is cognitively and emotionally inclined to accept, embrace, and adopt a particular plan to purposefully alter the status quo (Holt et al., 2007). Measured by - Readiness to Change Questionnaire (Revised Version) (RCQ) (Jakun version - to be validated). Outcomes can be pre-contemplation, contemplation, or action stage.
Motivation | 4 months
  An internal state or condition that activates behaviour and gives it direction (Edelman, 1997). Measured by Motivation Thought Frequency Scales for Alcohol (MTF-A) (Jakun version - to be validated). Higher MTF-A score implies higher motivation to quit or cut down alcohol use.
Self-efficacy | 4 months
  Individuals' beliefs or confidence in their capability to produce desired outcomes that affect their lives (Bandura & Wessels,1994). Measured by Brief Alcohol Abstinence Self-Efficacy 12-Item (AASE) Scale (Jakun version - to be validated). Higher AASE score indicates higher self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- RPS Kedaik & Kampung Jemeri, Kuala Rompin, Pahang, Malaysia

IPD SHARING:
Plan to Share IPD: No
Data will be securely retained for 7 years. Any disclosure of this information to a 3rd party will require explicit authorisation from MARA University of Technology, Malaysia.